CLINICAL TRIAL: NCT01793922
Title: A Prospective Randomized Multi-center Study Comparing Endoscopic Pneumodilation and Per Oral Endoscopic Myotomy (POEM) as Treatment of Idiopathic Achalasia
Brief Title: POEM Trial: Multi-center Study Comparing Endoscopic Pneumodilation and Per Oral Endoscopic Myotomy (POEM)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Guy Boeckxstaens, Prof. Dr., KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S55020
Record Dates: First submitted 2012-12-12; First posted 2013-02-18 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Achalasia
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PD (Active Comparator): pneumodilation
  Interventions: Procedure: PD
- POEM (Active Comparator): peroral endoscopic myotomy
  Interventions: Procedure: POEM

INTERVENTIONS:
Procedure: PD — pneumodilation
  Arms: PD
Procedure: POEM — peroral endoscopic myotomy
  Arms: POEM

SUMMARY:
The aim of the study is to compare the efficacy of per-oral endoscopic myotomy (POEM) to the efficacy of pneumodilation as the initial treatment of symptomatic idiopathic achalasia. It is hypothesized that POEM has a higher long-term efficacy than pneumodilation in treatment of therapy-naive patients with idiopathic achalasia.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 75 yr of age
* Manometric diagnosis of achalasia
* Eckardt score > 3
* Informed consent

Exclusion Criteria:

* Severe cardio-pulmonary disease or other serious disease leading to unacceptable surgical risk previous treatment, except treatment with nitroderivatives, Ca++ channel blockers or sildenafil, or dilation with Savary bougies or balloons of 2 cm diameter or smaller.

Pseudo-achalasia Mega-esophagus (> 7 cm) and/or sigmoid-like esophagus Previous esophageal or gastric surgery (except for gastric perforation) Not capable to fill out questionnaires (f.e. due to language barrier) Not available for follow-up Esophageal diverticula in the distal esophagus Malignant or premalignant esophageal lesions Patients with liver cirrhosis and/or esophageal varices Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-10; Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
therapeutic succes | 2 years
  The time till failure is the primary outcome parameter. The time is measured from date of pneumatic dilation (last session) or POEM to date of relapse of symptoms (date of establishment). Symptoms will be evaluated using the Eckardt scoring system (Table 1.). Therapeutic success is defined as a drop in Eckardt score to ≤ 3 after treatment and symptom control at yearly follow-up which is also defined as an Eckardt score of ≤ 3.
  If symptoms recur within patients randomized for pneumatic dilation, retreatment with pneumatic dilation is allowed according to the protocol. If retreatment does not result in reduction of the symptom score below 4, the patient will be considered as a treatment failure.

SECONDARY OUTCOMES:
quality of life | 2 years
  The quality of life is determined using a general QoL questionnaire, namely the SF36 questionnaire. In addition, a more disease specific questionnaire, i.e. the EORTC QLQ-OES24 questionnaire, is filled out. These questionnaires have scored the QoL at fixed time points during follow-up (1 month, 3 months and yearly).
complication rate | 2 years
  Complications (perforation, bleeding, etc) occurring during or immediately following the procedure are recorded by the attending phycisian.
  In addition, gastroesophageal reflux is measured using 24h pHmetry after 3 months and 1 year. The number of patients with pathological acid exposure (>4.5% of time a pH<4) will be assessed. Endoscopy is performed after 1 year to detect esophagitis. Esophagitis rates and LA grades of esophagitis will be assessed.
need for retreetment | 2 years
  Retreatment is allowed in the pneumodilation group when symptoms recur, which is defined as an Eckardt score of > 3. Symptom scores are assessed after one month, three months and then yearly.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium